CLINICAL TRIAL: NCT00133757
Title: Pharmacotherapy-assisted Extinction (Pharmacoextinction): A Novel Approach to the Treatment of Nicotine Dependence in Humans
Brief Title: Use of Pharmacotherapy to Reduce Cue-responsiveness in Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Peter Selby, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 114/2005
Record Dates: First submitted 2005-08-23; First posted 2005-08-24 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Nicotine Dependence; Tobacco Dependence
Keywords: Tobacco; Nicotine; Bupropion; Cue-reactivity; Craving
MeSH Terms: conditions — Tobacco Use Disorder

INTERVENTIONS:
Drug: Bupropion SR

SUMMARY:
In this study we, the investigators at the Centre for Addiction and Mental Health, intend to explore whether bupropion is able to reduce smokers' responses to cigarette-related environmental cues, and craving. Previous studies have indicated that bupropion may be able to achieve these outcomes. Therefore, we predict that smokers treated with bupropion for several weeks will show reduced reactivity to cigarette cues and craving.

DETAILED DESCRIPTION:
Current smoking cessation pharmacotherapy paradigms ignore the over-learned behaviour associated with smoking, thus contributing to the relatively poor absolute efficacy of pharmacotherapy. Chronic nicotine use causes adaptive changes in the brain that differ from the acute effects leading to craving when smoking is stopped. This is a key element of relapse. Thus, the development of more effective treatments involves a better understanding of craving and relapse by exploring the interaction between the psychology and neurobiology of nicotine addiction. Bupropion, an amphetamine derivative, has demonstrated efficacy in smoking cessation in motivated smokers. Its' mechanism of action is unclear but may be mediated by extinction processes. We hypothesize that bupropion will reduce cue-responsiveness and subsequent cravings in current smokers who are not consciously attempting to quit or cut down on smoking. Fifty smokers (>10 cigarettes/day) of either sex will be recruited to take either oral placebo or bupropion 150 mg twice daily for a total of 42 days. Subjects will attend bi-weekly experimental sessions where cue-responsiveness will be measured using physiological and subjective responses to a variety of neutral and smoking-related cues. Subjective effects will be measured using the Questionnaire of Smoking Urges, the Tobacco Craving Questionnaire and Visual Analog Scales. Subjects will record smoking behaviour and subjective experiences daily in a smoking diary. Outcome variables include cue responsiveness, daily diary ratings, exhaled end tidal CO levels, plasma cotinine levels, and subjective effects. Gender effects will be assessed by using sex as a covariate in the analysis. This study will provide preliminary data on pharmacotherapy-assisted extinction as a novel approach to smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* At least 19 years of age
* Smoking at least 10 cigarettes per day for at least 2 years
* Never treated with bupropion/Zyban

Exclusion Criteria:

* Co-morbid psychiatric disorder
* History of psychotic disorder or eating disorder
* Current alcohol or substance abuse/dependence (excluding nicotine, caffeine)
* Brain injury
* Seizure disorder
* Pregnancy, lactation, or at risk of becoming pregnant
* Current regular use of psychotropic drugs
* Known allergy or sensitivity to bupropion

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-06; Study Completion 2006-05

PRIMARY OUTCOMES:
Cue-responsiveness at pre, post, and during treatment
Craving at pre, post, and during treatment

SECONDARY OUTCOMES:
Attentional bias at pre and post treatment
Breath carbon monoxide levels at pre, post, and during treatment
Plasma cotinine levels at pre and post treatment
Puff topography measures at pre, post, and during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter Selby, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada